CLINICAL TRIAL: NCT02491684
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multi-centre Phase IIa Study in Asthma Patients Comparing the Efficacy and Safety of Once Daily Inhaled Interferon Beta-1a to Placebo, Administered for 14 Days After the Onset of Symptoms of an Upper Respiratory Tract Infection for the Prevention of Severe Exacerbations
Brief Title: A Study in Asthma Patients to Evaluate Efficacy, Safety and Tolerability of 14 Days Once Daily Inhaled Interferon Beta-1a After the Onset of Symptoms of an Upper Respiratory Tract Infection
Acronym: INEXAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D6230C00001
Record Dates: First submitted 2015-06-16; First posted 2015-07-08 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: asthma; Upper Respiratory Tract Infection; exacerbation; Interferon; efficacy; safety; prevention
MeSH Terms: conditions — Asthma; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (matching) (Placebo Comparator): Placebo, once daily inhalation for 14 days
  Interventions: Drug: Placebo
- Interferon beta-1a (Experimental): Interferon beta-1a, 24 μg (metered dose) once daily inhalation for 14 days
  Interventions: Drug: Interferon beta-1a Nebuliser solution 48 μg/mL

INTERVENTIONS:
Drug: Interferon beta-1a Nebuliser solution 48 μg/mL — Interferon beta-1a, 0,5 ml (24 μg, metered dose) once daily inhalation for 14 days
  Arms: Interferon beta-1a
Drug: Placebo — Placebo solution for once daily inhalation for 14 days
  Arms: Placebo (matching)

SUMMARY:
A study to investigate if inhaled Interferon beta-1a is safe and tolerated, and can prevent or reduce the severity of asthma attacks when administered to asthma patients at the onset of symptoms of common cold or influenza

DETAILED DESCRIPTION:
The study will consist of a Pre-Treatment Phase followed by a Treatment Phase. Patients are screened and enter the Pre-Treatment phase where they remain until they develop symptoms of a common cold or the flu. During this Pre-Treatment Phase patients will be asked daily if they think they have a common cold or the flu. When the patient answers yes to the question that he/she is coming down with a common cold or the flu, arrangements are made to evaluate the patient at the study site and, if eligible, enters the Treatment Phase. Baseline assessments are performed and the patient is randomized 1:1 to receive 24 μg (metered dose) inhaled Interferon beta-1a or placebo once daily for 14 days (delivered by the I-neb® device [Philips Respironics]). Treatment should start as soon as possible but no later than 48 hours after the onset of the first of the common cold or flu symptoms. Patients will be assessed with regards to exacerbations and changes in respiratory symptoms and reliever medication use at home using an ePRO device. Lung function will be measured both at home by the patients and at the study site. There will be five clinical visits during the Treatment Phase and two visits after the end of treatment; efficacy and safety will be monitored until 2-3 weeks after end of treatment when a final follow-up visit will take place.

The study population will comprise adult asthmatic patients on a maintenance treatment of medium to high dose inhaled corticosteroids and a second controller medication (eg, long- acting β2 agonist), with a documented history of at least two severe exacerbations within the last 24 months, of which at least one has occurred during the last 12 months, and it is suspected by the patient that these aforementioned exacerbations were triggered by an upper respiratory tract infection (ie, related to symptoms of a common cold or the flu).

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients should fulfil the following criteria:

1. Provision of signed and dated written informed consent prior to any study specific procedures
2. Male or female aged 18 and above at the time of enrolment
3. History of physician-diagnosed asthma requiring treatment with medium-to-high dose ICS (>250 μg fluticasone dry powder formulation equivalents total daily dose, as defined in GINA 2014, see CSP Appendix G), and a second controller medication as recommended in the GINA guidelines (ie, LABA, leukotriene receptor antagonist or sustained release theophylline). The medium or high dose ICS plus LABA can be any combination inhaler or 2 separate inhalers. Patients must have taken ICS (>250 μg fluticasone or the equivalent daily) plus second controller medication for at least 12 months prior to the date the informed consent is obtained, with or without another controller such as oral corticosteroids (OCS), theophylline, tiotropium, or leukotriene receptor antagonists. The maintenance treatment must have been kept at the same or at a higher level these last 12 months.
4. Proof of post-bronchodilator reversibility in FEV1 of ≥12% and ≥200 mL (Pellegrino et al 2005) documented within 5 years prior to Visit 1, or proof of a positive response to a methacholine or histamine challenge (a decrease in FEV1 by 20% [PC20] at ≤8 mg/mL) performed according to ATS/ERS guidelines (American Thoracic Society 2000) or proof of positive response to mannitol challenge (a decrease in FEV1 by 15% [PD15] at ≤635 mg) (Anderson et al 2009) documented within 5 years prior to Visit 1. If historical documentation is not available, reversibility or proof of a positive response to a methacholine, histamine or mannitol challenge must be demonstrated and documented at Visit 1
5. Must answer "Yes" to the question "Does a cold or flu make your asthma worse?"
6. To have had at least two documented severe asthma exacerbations within the last 24 months that were suspected by the patient to have been caused by a common cold or flu and To have had at least one documented severe asthma exacerbation within the last 12 months that was suspected by the patient to have been caused by a common cold or flu
7. Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception.
8. Negative pregnancy test (urine) for female patients of childbearing potential
9. Motivation (in the Investigator's opinion) to complete all study visits, the ability to communicate well with the Investigator and be capable of understanding the nature of the research and its treatment including its risks and benefits
10. Ability to read and write and use the electronic devices, including demonstrating an acceptable technique when using the ePRO device, home spirometer and the I-neb

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and staff at third party vendors or staff at the study sites)
2. Previous randomization to treatment in the present study
3. Any condition, including findings in the medical history or in the pre-study assessments that, in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the patient in the study or that could interfere with the study objectives, conduct or evaluation
4. Lung disease other than asthma (eg, chronic obstructive pulmonary disease, cystic fibrosis, allergic bronchopulmonary aspergillosis, active tuberculosis). Patients with CT or chest X-ray findings indicating bronchiectasis which in the opinion of the Investigator are not clinically significant may be enrolled at the discretion of the Investigator
5. Patients with ≥4 severe exacerbations during the last 12 months that the patient suspected were triggered by something else than an upper respiratory tract infection
6. Current participation in another clinical trial or participation in a clinical trial where the patient has received a dose of a test product (IMP) within 12 weeks prior to entry into the study for small molecules and within 12 months prior to entry into the study for biologicals, or 5 times the half-life (whichever is the longest) of the biologic or small molecule IMP
7. Patients who currently have, or have had within the past 3 months, any significant underlying medical condition(s) that could impact interpretation of results eg, infections, haematological disease, malignancy, renal, hepatic, coronary heart disease or other cardiovascular disease, including arrhythmias, endocrinological or gastrointestinal disease
8. Abnormal vital signs, after at least 10 minutes supine rest, defined as any of the following:

   * In patients < 60 years old, systolic blood pressure <90 mmHg or ≥150 mmHg
   * In patients ≥ 60 years old, systolic blood pressure <90 mmHg or ≥160 mmHg
   * Diastolic blood pressure <50 mmHg or ≥100 mmHg
   * HR <45 or >95 beats per minute
9. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, as considered by the Investigator, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology (particularly in the protocol defined primary lead) or left ventricular hypertrophy
10. Prolonged QTcF >450 ms (for both gender) or shortened QTcF <340 ms or family history of long QT syndrome
11. PR(PQ) interval shortening <120ms (PR<120 ms but >110 ms is acceptable if there is no evidence of ventricular pre-excitation).
12. PR(PQ) interval prolongation (>240ms), intermittent second or third degree AV block, or AV dissociation
13. QRS duration >120ms including persistent or intermittent bundle branch block
14. Patients with implantable cardiac defibrillator (ICD) or a permanent pacemaker and patients with symptomatic ventricular and / or atrial tachyarrhythmias
15. Patients with unstable angina pectoris or stable angina pectoris classified higher than Canadian Cardiovascular Society (CSS) class II or a myocardial infarction or stroke within 6 months
16. History of hospitalization within 12 months caused by heart failure or a diagnosis of heart failure higher than New York Heart Association (NYHA) class II
17. History of hypersensitivity to natural or recombinant Interferon beta-1a or to any of the drug preparation excipients
18. Received any marketed biologic agent (eg, omalizumab) within 12 months or 5 times the half-life (whichever is the longer) of the agent prior to enrolment
19. Significant history of depressive disorder or suicidal ideation. Specifically; individuals with current severe depression (ie, a low mood, which pervades all aspects of life and an inability to experience pleasure in activities that formerly were enjoyed); individuals with a past history of depression that required hospitalization or referral to psychiatric services in the past 5 years; individuals who currently feel suicidal or have attempted suicide in the past
20. History of epilepsy or seizures after the age of 5 years, other than febrile childhood seizure(s)
21. History of drug or alcohol abuse within 12 months prior to enrolment
22. Patients who have hepatic serum enzyme levels ≥2.5 times the normal range
23. Positive test for serum hepatitis B surface antigen, hepatitis C antibody, or HIV
24. Patients with a smoking history of ≥20 pack-years (1 pack year = 20 cigarettes smoked per day for one year)
25. Female who is breast-feeding, pregnant (verified by urine dipstick pregnancy test) or intends to become pregnant during the study
26. Patients who are unable to demonstrate an acceptable spirometry technique
27. Patients that have previously been included in studies evaluating the investigational medicinal product

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Gustafson, MD PhD, Study Director — AstraZeneca, R&D mölndal
Locations (32):
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonomade Buenos Aires
  - Research Site, Nueve de Julio
  - Research Site, Quilmes
- Australia (4):
  - Research Site, Bedford Park
  - Research Site, New Lambton
  - Research Site, Westmead
  - Research Site, Woolloongabba
- Colombia (2):
  - Research Site, Bogotá
  - Research Site, Floridablanca
- France (6):
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
- South Korea (3):
  - Research Site, Bucheon-si
  - Research Site, Jeonju
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Marbella (Málaga)
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (7):
  - Research Site, Blackpool
  - Research Site, Bradford
  - Research Site, Lancaster
  - Research Site, Leeds
  - Research Site, Manchester
  - Research Site, Nottingham
  - Research Site, Southampton

REFERENCES:
- [Derived] McCrae C, Olsson M, Gustafson P, Malmgren A, Aurell M, Fageras M, Da Silva CA, Cavallin A, Paraskos J, Karlsson K, Wingren C, Monk P, Marsden R, Harrison T. INEXAS: A Phase 2 Randomized Trial of On-demand Inhaled Interferon Beta-1a in Severe Asthmatics. Clin Exp Allergy. 2021 Feb;51(2):273-283. doi: 10.1111/cea.13765. Epub 2020 Nov 3. PMID 33091192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 21 July 2015; Last Patient Last Visit: 24 November 2016. The study was performed at 39 sites in 7 countries including Argentina, Australia, Colombia, France, South Korea, Spain and the United Kingdom.
Pre-assignment Details: 349 patients enrolled (signed informed consent) and 228 were not randomised. 121 patients met randomisation criteria and entered the pre-treatment phase. Patients were treated after developing symptoms of an upper respiratory tract infection (URTI) if they met all the inclusion criteria and none of the exclusion criteria for the treatment phase.
Groups:
- AZD9412: Patients were randomised to receive investigational product AZD9412 (interferon beta-1a) in the treatment phase.
  Eligible patients entered the pre-treatment phase until they developed symptoms of a common cold or flu (URTI). Patients were evaluated at a study site for eligibility to enter the treatment phase as soon as possible but no later than 48 hours after the onset of the first symptoms of an URTI.
  Patients randomised to the AZD9412 group received 6 Million International Units (MIU) (24 micrograms [mcg] metered dose) inhaled AZD9412 once daily for 14 days, delivered by the I-neb® device.
  Patients continued their regular asthma maintenance treatment, and were assessed for exacerbations, changes in respiratory symptoms and reliever medication use using an electronic Patient Reported Outcome (ePRO) device at home.
- Placebo: Patients were randomised to receive placebo in the treatment phase. Eligible patients entered the pre-treatment phase until they developed symptoms of a common cold or the flu (URTI). Patients were evaluated at a study site for eligibility to enter the treatment phase as soon as possible but no later than 48 hours after the onset of the first symptoms of an URTI.
  Patients randomised to the placebo group received 6 MIU (24 mcg metered dose) inhaled placebo once daily for 14 days, delivered by the I-neb® device.
  Patients continued their regular asthma maintenance treatment, and were assessed for exacerbations, changes in respiratory symptoms and reliever medication use using an ePRO device at home.
Period: Pre-treatment Phase
Arm/Group | AZD9412 | Placebo
Started | 61 | 60
Completed | 61 | 60
Not Completed | 0 | 0
Period: Treatment Phase
Arm/Group | AZD9412 | Placebo
Started | 61 | 60
Completed | 58 | 57
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Incorrect randomisation | 1 | 0
Not completed — Investigator and Sponsor decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- AZD9412: Patients were randomised to receive investigational product AZD9412 (interferon beta-1a) in the treatment phase.
  Eligible patients entered the pre-treatment phase until they developed symptoms of a common cold or flu (URTI). Patients were evaluated at a study site for eligibility to enter the treatment phase as soon as possible but no later than 48 hours after the onset of the first symptoms of an URTI.
  Patients randomised to the AZD9412 group received 6 MIU (24 mcg metered dose) inhaled AZD9412 once daily for 14 days, delivered by the I-neb® device.
  Patients continued their regular asthma maintenance treatment, and were assessed for exacerbations, changes in respiratory symptoms and reliever medication use using an ePRO device at home.
- Total: Total of all reporting groups
Arm/Group | AZD9412 | Placebo | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.95) | 47.7 (14.10) | 47.7 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 43 | 91
  Male | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Severe Asthma Exacerbation During 14 Days of Treatment
Description: Evaluation of the efficacy of inhaled AZD9412 compared to placebo in preventing severe exacerbations during the 14 day treatment phase following the onset of an URTI in asthmatic patients.
  A severe exacerbation was defined as worsening asthma symptoms and
  1. use of systemic corticosteroids (or a temporary increase of at least 2-fold in a stable oral corticosteroid background dose) for at least 3 consecutive days and/or
  2. an unscheduled visit or emergency room visit due to asthma symptoms that required at least 1 dose of systemic corticosteroids and/or
  3. an in-patient hospitalisation due to asthma requiring at least 1 dose of systemic corticosteroids.
  The number of patients with severe asthma exacerbations with onset during the treatment phase is presented for each treatment group.
Time Frame: Day 1 - 14 of the treatment phase.
Population: The Intention to treat (ITT) analysis set consisted of all randomised patients who received at least 1 dose of investigational product and had some post-dose data available.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Participants | 7 | 5
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Proportions of patients with exacerbations are compared using a log-binomial regression model with treatment group and region as factors; Test type: Superiority or Other; p = 0.645, log-binomial regression model; The ratio of proportions was calculated by back-transforming the estimated treatment effect; Ratio of proportions = 1.29, 95% CI 2-sided [0.43 to 3.85] — AZD9412 versus Placebo

2. Secondary Outcome: Proportion of Patients With Severe Asthma Exacerbations Within 7 and 30 Days Following Randomisation
Description: Evaluation of the efficacy of inhaled AZD9412 compared to placebo in preventing severe exacerbations within 7 and 30 days after the start of treatment (Day 1).
  A severe exacerbation was defined as worsening asthma symptoms and
  1. use of systemic corticosteroids (or a temporary increase of at least 2-fold in a stable oral corticosteroid background dose) for at least 3 consecutive days and/or
  2. an unscheduled visit or emergency room visit due to asthma symptoms that required at least 1 dose of systemic corticosteroids and/or
  3. an in-patient hospitalisation due to asthma requiring at least 1 dose of systemic corticosteroids.
  The numbers of patients with severe asthma exacerbations with onset during Days 1 - 7 and Days 1 - 30 are presented for each treatment group.
Time Frame: Day 1 of treatment phase up to 30 days post-randomisation.
Population: The ITT analysis set consisted of all randomised patients who received at least 1 dose of investigational product and had some post-dose data available.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Participants
  Days 1 - 7 | 4 | 2
  Days 1 - 30 | 8 | 6
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.411, log-binomial regression model; The ratio of proportions was calculated by back-transforming the estimated treatment effect; Ratio of proportions = 1.97, 95% CI 2-sided [0.39 to 9.89] — AZD9412 versus Placebo for Days 1 - 7
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.659, log-binomial regression model; The ratio of proportions was calculated by back-transforming the estimated treatment effect; Ratio of proportions = 1.25, 95% CI 2-sided [0.46 to 3.41] — AZD9412 versus Placebo for Days 1 - 30

3. Secondary Outcome: Proportion of Patients With Moderate Asthma Exacerbation Within 7, 14 and 30 Days Following Randomisation
Description: Evaluation of the efficacy of inhaled AZD9412 compared to placebo in preventing moderate exacerbations within 7, 14 and 30 days after the start of treatment (Day 1).
  A moderate exacerbation was defined as a temporary increase in maintenance therapy in order to prevent a severe event supported by a sustained (2 or more days) worsening in at least one key control metric, including asthma score, rescue use, night time awakening or morning peak expiratory flow.
  The numbers of patients with moderate exacerbations with onset during Days 1 - 7, Days 1 - 14 and Days 1 - 30 are presented for each treatment group.
  With respect to the Day 1-7 analysis, the model did not converge so the analysis could not be performed.
Time Frame: Day 1 of treatment phase up to 30 days post-randomisation.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Participants
  Days 1 - 7 | 0 | 1
  Days 1 - 14 | 1 | 1
  Days 1 - 30 | 1 | 1
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.944, log-binomial regression model; The ratio of proportions was calculated by back-transforming the estimated treatment effect; Ratio of proportions = 1.10, 95% CI 2-sided [0.08 to 15.79] — AZD9412 versus Placebo for Days 1 - 14
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.944, log-binomial regression model; The ratio of proportions was calculated by back-transforming the estimated treatment effect; Ratio of proportions = 1.10, 95% CI 2-sided [0.08 to 15.79] — AZD9412 versus Placebo for Days 1 - 30

4. Secondary Outcome: Time to First Severe Asthma Exacerbation During 30 Days Following Randomisation
Description: The time to first event was calculated as start date of events - date of randomisation + 1.
  Patients with no observed event were censored at the date of their last visit, or for lost-to-follow-up patients, at the last time point after which an event could not be assessed.
  The median time to first exacerbation was not calculated in either treatment group due to low numbers of events.
Time Frame: From Day 1 of treatment phase up to 30 days post-randomisation.
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Days | NA [NA to NA] — The median time to severe exacerbation was not calculated due to low numbers of events. | NA [NA to NA] — The median time to severe exacerbation was not calculated due to low numbers of events.
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of time to first severe exacerbation within 30 days of treatment start; Test type: Superiority or Other; p = 0.634, Regression, Cox; Hazard ratio was calculated adjusting for treatment group and region; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.45 to 3.77] — AZD9412 versus Placebo

5. Secondary Outcome: Time to First Moderate Asthma Exacerbation During 30 Days Following Randomisation
Description: as for outcome 4
Time Frame: From Day 1 of treatment phase up to 30 days post-randomisation.
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Days | NA [NA to NA] — The median time to moderate exacerbation was not calculated due to low numbers of events. | NA [NA to NA] — The median time to moderate exacerbation was not calculated due to low numbers of events.
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of time to first moderate exacerbation within 30 days of treatment start; Test type: Superiority or Other; p = 0.973, Regression, Cox; Hazard ratio was calculated adjusting for treatment group and region; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.07 to 16.78] — AZD9412 versus Placebo

6. Secondary Outcome: Duration of Moderate or Severe Exacerbations
Description: The duration of each individual moderate or severe exacerbation was calculated as:
  Cessation date of exacerbation - Start date of exacerbation + 1.
  The start date of a severe exacerbation was defined as the start date of systemic corticosteroids or increase of systemic corticosteroids or emergency room visit or hospital admission, whichever occurred first. The stop date was defined as the last day of systemic corticosteroids/increase of systemic corticosteroids or hospital discharge, whichever occurred last.
  The start date of a moderate exacerbation was defined as the first day of increase in temporary maintenance therapy. The stop date was defined as the last day of this treatment.
  The mean duration of moderate or severe exacerbations is presented for each treatment group.
Time Frame: Day 1 of treatment phase up to 30 days post-randomisation.
Population: The ITT analysis set consisted of all randomised patients who received at least 1 dose of investigational product and had some post-dose data available.
  The number of patients in the analysis are those with at least 1 exacerbation.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 8 | 6
Days | 10 (7.7) | 8 (4.5)

7. Secondary Outcome: Change in Asthma Control From Baseline up to 30 Days as Measured by the Asthma Control Questionnaire (ACQ-6)
Description: The ACQ-6 consists of 6 questions to assess asthma control, each question measured on a 7-point scale scored from 0 (totally controlled) to 6 (severely uncontrolled). The ACQ-6 total score is computed as the un-weighted mean of the responses to the 6 questions. Baseline assessments were taken as the last non-missing assessment prior to randomisation.
  The change from baseline at Visit 4 (Day 7 +/- 1), at Visit 6 (Day 14 +/- 1) and at Visit 8 (Day 30) is presented for the total score and for each of the 6 questions.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: The ITT analysis set consisted of all randomised patients who received at least 1 dose of investigational product and had some post-dose data available.
  Patients with non-missing values were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Units on a Scale
  ACQ-6 Total Score, Visit 4: number analyzed (Participants) | 53 | 54
  ACQ-6 Total Score, Visit 4 | 0.02 (0.11) | -0.07 (0.12)
  ACQ-6 Total Score, Visit 6: number analyzed (Participants) | 57 | 55
  ACQ-6 Total Score, Visit 6 | -0.15 (0.14) | -0.21 (0.14)
  ACQ-6 Total Score, Visit 8: number analyzed (Participants) | 55 | 56
  ACQ-6 Total Score, Visit 8 | -0.42 (0.15) | -0.35 (0.15)
  Q1: Woken by Asthma, Visit 4: number analyzed (Participants) | 53 | 54
  Q1: Woken by Asthma, Visit 4 | 0.09 (0.18) | -0.09 (0.18)
  Q1: Woken by Asthma, Visit 6: number analyzed (Participants) | 57 | 55
  Q1: Woken by Asthma, Visit 6 | 0.15 (0.20) | -0.28 (0.21)
  Q1: Woken by Asthma, Visit 8: number analyzed (Participants) | 55 | 56
  Q1: Woken by Asthma, Visit 8 | -0.50 (0.18) | -0.32 (0.18)
  Q2: Symptoms at Awakening, Visit 4: number analyzed (Participants) | 53 | 54
  Q2: Symptoms at Awakening, Visit 4 | 0.06 (0.18) | -0.17 (0.18)
  Q2: Symptoms at Awakening, Visit 6: number analyzed (Participants) | 57 | 55
  Q2: Symptoms at Awakening, Visit 6 | -0.40 (0.16) | -0.33 (0.17)
  Q2: Symptoms at Awakening, Visit 8: number analyzed (Participants) | 55 | 56
  Q2: Symptoms at Awakening, Visit 8 | -0.76 (0.19) | -0.47 (0.19)
  Q3: Limited in Activities, Visit 4: number analyzed (Participants) | 53 | 54
  Q3: Limited in Activities, Visit 4 | 0.04 (0.15) | 0.06 (0.15)
  Q3: Limited in Activities, Visit 6: number analyzed (Participants) | 57 | 55
  Q3: Limited in Activities, Visit 6 | -0.12 (0.17) | 0.16 (0.18)
  Q3: Limited in Activities, Visit 8: number analyzed (Participants) | 55 | 56
  Q3: Limited in Activities, Visit 8 | -0.43 (0.18) | -0.33 (0.18)
  Q4: Shortness of Breath, Visit 4: number analyzed (Participants) | 53 | 54
  Q4: Shortness of Breath, Visit 4 | -0.13 (0.15) | -0.11 (0.16)
  Q4: Shortness of Breath, Visit 6: number analyzed (Participants) | 57 | 55
  Q4: Shortness of Breath, Visit 6 | -0.34 (0.19) | -0.38 (0.21)
  Q4: Shortness of Breath, Visit 8: number analyzed (Participants) | 55 | 56
  Q4: Shortness of Breath, Visit 8 | -0.46 (0.18) | -0.37 (0.19)
  Q5: Wheeze, Visit 4: number analyzed (Participants) | 53 | 54
  Q5: Wheeze, Visit 4 | 0.13 (0.17) | 0.08 (0.17)
  Q5: Wheeze, Visit 6: number analyzed (Participants) | 57 | 55
  Q5: Wheeze, Visit 6 | -0.17 (0.17) | -0.17 (0.18)
  Q5: Wheeze, Visit 8: number analyzed (Participants) | 55 | 56
  Q5: Wheeze, Visit 8 | -0.33 (0.21) | -0.42 (0.21)
  Q6: Puffs of Short-Acting Bronchodilator; Visit 4: number analyzed (Participants) | 53 | 54
  Q6: Puffs of Short-Acting Bronchodilator; Visit 4 | 0.06 (0.13) | 0.00 (0.14)
  Q6: Puffs of Short-Acting Bronchodilator; Visit 6: number analyzed (Participants) | 57 | 55
  Q6: Puffs of Short-Acting Bronchodilator; Visit 6 | 0.07 (0.14) | -0.11 (0.15)
  Q6: Puffs of Short-Acting Bronchodilator; Visit 8: number analyzed (Participants) | 55 | 56
  Q6: Puffs of Short-Acting Bronchodilator; Visit 8 | 0.04 (0.14) | -0.03 (0.14)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of change from baseline in total score at Visit 4; Test type: Superiority or Other; p = 0.495, ANCOVA; Change from baseline is analysed using an Analysis of Covariance (ANCOVA) model with treatment and region as factors and baseline value as covariate; Least Squares (LS) Mean difference = 0.09, 95% CI 2-sided [-0.17 to 0.35] — AZD9412 versus Placebo for change from baseline in total score at Visit 4
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; Analysis of change from baseline in total score at Visit 6; Test type: Superiority or Other; p = 0.715, ANCOVA; Change from baseline is analysed using an ANCOVA model with treatment and region as factors and baseline value as covariate; LS Mean Difference = 0.06, 95% CI 2-sided [-0.26 to 0.38] — AZD9412 versus Placebo
Statistical Analysis 3: Comparison: AZD9412 vs Placebo; Analysis of change from baseline in total score at Visit 8; Test type: Superiority or Other; p = 0.687, ANCOVA; [statistical method as in outcome 7, analysis 2]; LS Mean Difference = -0.07, 95% CI 2-sided [-0.42 to 0.28] — AZD9412 versus Placebo

8. Secondary Outcome: AUC for Change in Daytime and Night-time Asthma Symptom Score From Baseline up to 30 Days
Description: Asthma symptoms during night-time and daytime were recorded by the patient each morning and evening in the Asthma Daily Diary on a daily basis. Symptoms were recorded using a scale of 0 to 3 where 0 indicates no asthma symptoms up to an absolute score of 3. Baseline assessments were taken as the last non-missing assessment prior to randomisation. The total daily asthma symptom score was calculated by taking the sum of the night-time and daytime asthma scores recorded each day. The outcome variable is the area under the curve (AUC) for change from baseline in day-time, night-time and total daily asthma symptom scores over Days 1-14, Days 1-7, Days 8-14 and Days 15-30.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on Scale
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Units on Scale
  Total asthma score, Days 1-14: number analyzed (Participants) | 47 | 46
  Total asthma score, Days 1-14 | -0.20 (0.16) | -0.31 (0.16)
  Total asthma score, Days 1-7: number analyzed (Participants) | 48 | 50
  Total asthma score, Days 1-7 | -0.11 (0.13) | -0.22 (0.13)
  Total asthma score, Days 8-14: number analyzed (Participants) | 54 | 49
  Total asthma score, Days 8-14 | -0.40 (0.15) | -0.41 (0.16)
  Total asthma score, Days 15-30: number analyzed (Participants) | 55 | 55
  Total asthma score, Days 15-30 | -0.77 (0.16) | -0.77 (0.16)
  Daytime asthma score, Days 1-14: number analyzed (Participants) | 56 | 56
  Daytime asthma score, Days 1-14 | -0.22 (0.07) | -0.26 (0.07)
  Daytime asthma score, Days 1-7: number analyzed (Participants) | 56 | 58
  Daytime asthma score, Days 1-7 | -0.17 (0.06) | -0.17 (0.06)
  Daytime asthma score, Days 8-14: number analyzed (Participants) | 58 | 57
  Daytime asthma score, Days 8-14 | -0.23 (0.07) | -0.27 (0.07)
  Daytime asthma score, Days 15-30: number analyzed (Participants) | 60 | 59
  Daytime asthma score, Days 15-30 | -0.44 (0.07) | -0.41 (0.07)
  Night-time asthma score, Days 1-14: number analyzed (Participants) | 53 | 50
  Night-time asthma score, Days 1-14 | -0.17 (0.07) | -0.16 (0.08)
  Night-time asthma score, Days 1-7: number analyzed (Participants) | 54 | 52
  Night-time asthma score, Days 1-7 | -0.10 (0.06) | -0.09 (0.07)
  Night-time asthma score, Days 8-14: number analyzed (Participants) | 55 | 53
  Night-time asthma score, Days 8-14 | -0.20 (0.07) | -0.17 (0.08)
  Night-time asthma score, Days 15-30: number analyzed (Participants) | 57 | 55
  Night-time asthma score, Days 15-30 | -0.44 (0.09) | -0.39 (0.09)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline in total score over Days 1-14; Test type: Superiority or Other; p = 0.516, ANCOVA; AUC for change from baseline is analysed using an ANCOVA model with treatment and region as factors and baseline value as covariate; LS Mean difference = 0.11, 95% CI 2-sided [-0.23 to 0.45] — AZD9412 versus Placebo
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline in total score over Days 1-7; Test type: Superiority or Other; p = 0.417, ANCOVA; [statistical method as in outcome 8, analysis 1]; LS mean difference = 0.11, 95% CI 2-sided [-0.16 to 0.37] — AZD9412 versus Placebo
Statistical Analysis 3: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline in total score over Days 8-14; Test type: Superiority or Other; p = 0.954, ANCOVA; [statistical method as in outcome 8, analysis 1]; LS mean difference = 0.01, 95% CI 2-sided [-0.34 to 0.36] — AZD9412 versus Placebo
Statistical Analysis 4: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline in total score over Days 15-30; Test type: Superiority or Other; p = 0.985, ANCOVA; [statistical method as in outcome 8, analysis 1]; LS Mean difference = 0.00, 95% CI 2-sided [-0.35 to 0.35] — AZD9412 versus Placebo

9. Secondary Outcome: Change in the Proportion of Night-time Awakening Using the ePRO Questionnaire From Baseline up to 30 Days
Description: Night-time awakenings due to asthma symptoms were recorded by the patient in the Asthma Daily Diary each morning by answering the question whether he/she woke up during the night due to asthma symptoms with a 'yes' or 'no' response.
  Biweekly means were calculated as the percentages of times the subject answered 'yes' over a period of 14 sequential days. Biweekly means are presented for the periods over Days 2-15 and Days 16-30.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of 'yes' responses
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Percentage of 'yes' responses
  Days 2-15 | 22.3 (30.42) | 24.8 (29.77)
  Days 16-30: number analyzed (Participants) | 60 | 59
  Days 16-30 | 15.2 (26.79) | 15.9 (26.34)

10. Secondary Outcome: Change in Health-related Quality of Life as Measured by the Asthma Quality of Life Questionnaire (AQLQ[S]) From Baseline up to 30 Days
Description: The AQLQ(S) was used to assess health-related quality of life and consisted of 32 questions. Patients were asked to score each of the questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The questions were allocated to 4 domains assessing:
  1. activity limitation,
  2. symptoms,
  3. emotional function, and
  4. environmental stimuli
  The overall score was calculated as the mean of the responses to all questions. The mean change in overall score from baseline at Visit 6 (Day 14+/-1) and Visit 8 (Day 30) are presented.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on Scale
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
Units on Scale
  Overall Score Visit 6: number analyzed (Participants) | 57 | 56
  Overall Score Visit 6 | 0.28 (0.13) | 0.35 (0.14)
  Overall Score Visit 8: number analyzed (Participants) | 55 | 57
  Overall Score Visit 8 | 0.43 (0.16) | 0.53 (0.16)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of change from baseline in overall score at Visit 6; Test type: Superiority or Other; p = 0.660, ANCOVA; [statistical method as in outcome 7, analysis 2]; LS Mean difference = -0.07, 95% CI 2-sided [-0.38 to 0.24] — AZD9412 versus Placebo
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; Analysis of change from baseline in overall score at Visit 8; Test type: Superiority or Other; p = 0.624, ANCOVA; [statistical method as in outcome 7, analysis 2]; LS Mean difference = -0.09, 95% CI 2-sided [-0.48 to 0.29] — AZD9412 versus Placebo

11. Secondary Outcome: AUC for Change in Daytime and Night-time Reliever Medication Use From Baseline up to 14 Days
Description: Patients recorded the number of reliever medication inhalations taken twice daily in the Asthma Daily Diary. The number of inhalations taken between the morning and evening lung function assessments were recorded in the evening. The number of inhalations taken between the evening and morning lung function assessments were recorded in the morning. Baseline assessments were taken as the last non-missing assessment prior to randomisation.
  The AUC for change from baseline over Days 1-14 (inclusive of Days 1 and 14) is presented.
Time Frame: From baseline up to Day 14 of treatment phase.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Inhalations
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 52 | 48
Inhalations | -0.12 (0.46) | -0.67 (0.48)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-14; Test type: Superiority or Other; p = 0.309, ANCOVA; [statistical method as in outcome 8, analysis 1]; LS Mean difference = 0.54, 95% CI 2-sided [-0.51 to 1.59] — AZD9412 versus Placebo

12. Secondary Outcome: AUC for Change in the Morning Peak Expiratory Flow (PEF) From Baseline to up to 30 Days
Description: Patients measured morning PEF at home and recorded the results using the ePRO device. Baseline assessments were taken as the last non-missing assessment prior to randomisation.
  The mean AUC for change from baseline is presented for the periods Days 1-14, 1-7, 8-14 and 15-30.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: litres/minute (l/min)
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
litres/minute (l/min)
  Days 1-14: number analyzed (Participants) | 55 | 57
  Days 1-14 | 9.56 (14.02) | -7.42 (13.91)
  Days 1-7: number analyzed (Participants) | 56 | 59
  Days 1-7 | 19.66 (9.66) | 0.31 (9.11)
  Days 8-14: number analyzed (Participants) | 57 | 57
  Days 8-14 | 7.03 (15.90) | -7.35 (15.80)
  Days 15-30: number analyzed (Participants) | 59 | 59
  Days 15-30 | 32.75 (15.35) | 13.49 (14.82)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-14; Test type: Superiority or Other; p = 0.059, ANCOVA; Analysis uses an ANCOVA model with treatment, region, gender, and smoking status as factors, and baseline value and height as covariates; LS Mean difference = 16.98, 95% CI 2-sided [-0.63 to 34.60] — AZD9412 versus Placebo
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-7; Test type: Superiority or Other; p = 0.010, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 19.35, 95% CI 2-sided [4.66 to 34.05] — AZD9412 versus Placebo
Statistical Analysis 3: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 8-14; Test type: Superiority or Other; p = 0.153, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 14.38, 95% CI 2-sided [-5.44 to 34.20] — AZD9412 versus Placebo
Statistical Analysis 4: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 15-30; Test type: Superiority or Other; p = 0.096, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 19.26, 95% CI 2-sided [-3.44 to 41.97] — AZD9412 versus Placebo

13. Secondary Outcome: AUC for Change in the Morning Forced Expiratory Volume in 1 Second (FEV1) From Baseline up to 30 Days
Description: Patients measured morning FEV1 at home and recorded the results using the ePRO device. Baseline assessments were taken as the last non-missing assessment prior to randomisation.
  The mean AUC for change from baseline is presented for the periods Days 1-14, 1-7, 8-14 and 15-30.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
litres
  Days 1-14: number analyzed (Participants) | 55 | 57
  Days 1-14 | -0.00 (0.08) | -0.08 (0.08)
  Days 1-7: number analyzed (Participants) | 56 | 59
  Days 1-7 | 0.10 (0.06) | 0.02 (0.06)
  Days 8-14: number analyzed (Participants) | 57 | 57
  Days 8-14 | -0.03 (0.08) | -0.09 (0.08)
  Days 15-30: number analyzed (Participants) | 59 | 59
  Days 15-30 | 0.15 (0.09) | 0.04 (0.08)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-14; Test type: Superiority or Other; p = 0.161, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.07, 95% CI 2-sided [-0.03 to 0.17] — AZD9412 versus Placebo
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-7; Test type: Superiority or Other; p = 0.087, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.08, 95% CI 2-sided [-0.01 to 0.17] — AZD9412 versus Placebo
Statistical Analysis 3: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 8-14; Test type: Superiority or Other; p = 0.280, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.16] — AZD9412 versus Placebo
Statistical Analysis 4: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 15-30; Test type: Superiority or Other; p = 0.086, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.11, 95% CI 2-sided [-0.02 to 0.24] — AZD9412 versus Placebo

14. Secondary Outcome: AUC for Change in the Evening PEF From Baseline to up to 30 Days
Description: Patients measured evening PEF at home and recorded the results using the ePRO device. Baseline assessments were taken as the last non-missing assessment prior to randomisation.
  The mean AUC for change from baseline is presented for the periods Days 1-14, 1-7, 8-14 and 15-30.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: l/min
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
l/min
  Days 1-14: number analyzed (Participants) | 52 | 51
  Days 1-14 | 10.96 (12.58) | -0.73 (11.88)
  Days 1-7: number analyzed (Participants) | 53 | 53
  Days 1-7 | 8.78 (9.87) | -2.41 (9.30)
  Days 8-14: number analyzed (Participants) | 53 | 52
  Days 8-14 | 8.49 (13.09) | -2.66 (12.55)
  Days 15-30: number analyzed (Participants) | 56 | 54
  Days 15-30 | 11.88 (15.70) | -5.25 (15.13)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-14; Test type: Superiority or Other; p = 0.211, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 11.69, 95% CI 2-sided [-6.76 to 30.14] — AZD9412 versus Placebo
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-7; Test type: Superiority or Other; p = 0.125, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 11.19, 95% CI 2-sided [-3.18 to 25.56] — AZD9412 versus Placebo
Statistical Analysis 3: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 8-14; Test type: Superiority or Other; p = 0.277, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 11.14, 95% CI 2-sided [-9.08 to 31.36] — AZD9412 versus Placebo
Statistical Analysis 4: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 15-30; Test type: Superiority or Other; p = 0.161, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 17.13, 95% CI 2-sided [-6.92 to 41.18] — AZD9412 versus Placebo

15. Secondary Outcome: AUC for Change in the Evening FEV1 From Baseline up to 30 Days
Description: Patients measured evening FEV1 at home and recorded the results using the ePRO device. Baseline assessments were taken as the last non-missing assessment prior to randomisation.
  The mean AUC for change from baseline is presented for the periods Days 1-14, 1-7, 8-14 and 15-30.
Time Frame: From baseline up to 30 days after start of treatment phase.
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | AZD9412 | Placebo
Number analyzed (Participants) | 61 | 60
litres
  Days 1-14: number analyzed (Participants) | 52 | 51
  Days 1-14 | -0.01 (0.07) | -0.07 (0.07)
  Days 1-7: number analyzed (Participants) | 53 | 53
  Days 1-7 | 0.01 (0.07) | -0.03 (0.07)
  Days 8-14: number analyzed (Participants) | 53 | 52
  Days 8-14 | -0.02 (0.07) | -0.08 (0.07)
  Days 15-30: number analyzed (Participants) | 56 | 54
  Days 15-30 | 0.02 (0.08) | -0.08 (0.08)
Statistical Analysis 1: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-14; Test type: Superiority or Other; p = 0.287, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.06, 95% CI 2-sided [-0.05 to 0.16] — AZD9412 versus Placebo
Statistical Analysis 2: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 1-7; Test type: Superiority or Other; p = 0.457, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.04, 95% CI 2-sided [-0.06 to 0.14] — AZD9412 versus Placebo
Statistical Analysis 3: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 8-14; Test type: Superiority or Other; p = 0.315, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.05, 95% CI 2-sided [-0.05 to 0.16] — AZD9412 versus Placebo
Statistical Analysis 4: Comparison: AZD9412 vs Placebo; Analysis of AUC for change from baseline over Days 15-30; Test type: Superiority or Other; p = 0.134, ANCOVA; [statistical method as in outcome 12, analysis 1]; LS Mean difference = 0.09, 95% CI 2-sided [-0.03 to 0.22] — AZD9412 versus Placebo

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from the first day of study treatment up to the last date of follow-up (approximately 30 days).
Description: The safety analysis set consisted of all randomised patients who received at least 1 dose of investigational product and with post-dose data available.
Arm/Group | AZD9412 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/61 | 0/60
Other Adverse Events (participants affected / at risk) | 27/61 | 20/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9412 (N=61) | Placebo (N=60)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9412 (N=61) | Placebo (N=60)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (3) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injury associated with device (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to the lower than expected rate of severe exacerbations in the study as a whole, and due to the observed lack of differential effect at interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other